CLINICAL TRIAL: NCT01281501
Title: A Randomized, Controlled Trial of Adding Intravenous Pantoprazole to Conventional Treatment for the Immediate Relief of Dyspeptic Pain
Brief Title: Symptomatic Relief of Acute Dyspeptic Pain in Emergency Department With Pantoprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khrongwong Musikatavorn, MD., Department of Medicine, Faculty of Medicine, Chulalongkorn University and King Chulalongkorn Memorial Hospital., Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 619/2010
Record Dates: First submitted 2011-01-17; First posted 2011-01-24 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Dyspepsia; Emergency; Pain
Keywords: Dyspepsia; Emergency treatment; Pantoprazole; Antacid; Pain measurement
MeSH Terms: conditions — Dyspepsia; Emergencies; Pain | interventions — Saline Solution; Pantoprazole; Antacids; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional (Active Comparator): Oral antacid, 20 mg of intravenous hyoscine butylbromide, normal saline
  Interventions: Drug: Normal saline; Drug: Oral antacid; Drug: Hyoscine butylbromide
- Pantoprazole (Experimental): Oral antacid, 20 mg of intravenous hyoscine butylbromide, 80 mg of intravenous pantoprazole
  Interventions: Drug: Pantoprazole; Drug: Oral antacid; Drug: Hyoscine butylbromide

INTERVENTIONS:
Drug: Normal saline — 10 ml of 0.9% sodium chloride solution
  Arms: Conventional
Drug: Pantoprazole — 80 mg of intravenous pantoprazole
  Other Names: Controloc (Protonix)
  Arms: Pantoprazole
Drug: Oral antacid — 30 ml of oral antacid (1.32 grams of aluminum hydroxide, 0.72 grams of magnesium hydroxide)
  Other Names: Antacid
Drug: Hyoscine butylbromide — 20 mg of intravenous hyoscine butylbromide
  Other Names: Buscopan

SUMMARY:
The purpose of this study is to evaluate the immediate synergistic effect on the relief of severe acid-related dyspeptic pain by adding intravenous pantoprazole to the combination of oral antacid and antispasmodic agent (the conventional treatment).

DETAILED DESCRIPTION:
Acid-related dyspepsia is common among the population. Number of these patients may have so severe symptoms that can lead them to the emergency department. Mixtures of antacid and antispasmodic were widely used over decades to relieve this acute pain with moderate, yet questionable, improvement in pain score. Proton pump inhibitors (PPIs), the novel acid-lowering agents, are undoubtedly effective to reduce acid secretion and control dyspeptic symptoms in short-term and long-term duration. To our knowledge, no previous study was conducted to evaluate the efficacy of such agents on immediate pain relief in patients with severe dyspeptic symptoms in emergency care. Clinically, they are frequently used to treat this circumstance in an unofficial manner since intravenous proton pump inhibitor alone is not yet considered as a well-approved indication to alleviate such condition. Pantoprazole, a proton pump inhibitor, reaches its peak serum concentration within one hour and its acid-lowering effect occurred within first hour following a single intravenous infusion. Thus, it theoretically has rapid onset and prolonged action on acid reduction. Our primary aim of the study is to evaluate the immediate effect of intravenous pantoprazole in addition to the combination of oral antacid and antispasmodic agent (the conventional regimen) on the relief of severe acid-related dyspeptic pain.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acid-related dyspepsia
* age 15 to 50 years

Exclusion Criteria:

* pre-treatment 100-millimeter linear Visual Analog Scale (100-mm VAS) pain scores less than 5.0
* known cases of malignancies or terminal illnesses
* known cases of major medical problems
* allergic to studied drugs
* contraindicated to hyoscine butylbromide (glaucoma, myasthenia gravis, paralytic ileus, pyloric stenosis, prostatic enlargement, porphyria)
* received acid antisecretory agents (proton pump inhibitors or histamine-2 receptor antagonists), antispasmodic agents, alcoholic consumption, nonsteroidal anti-inflammatory drugs, aspirin and steroids within 5 days or oral antacids within 4 hours prior to the visit
* receiving clopidogrel, statins, iron therapies, warfarins, antiretroviral agents, which may have serious drug interaction with the proton pump inhibitors
* receiving drugs that have strong anticholinergic activities (e.g. acetylcholinesterase inhibitors for Parkinson's or Alzheimer diseases, antihistamines, antispasmodic agents, antipsychotics, skeletal muscle relaxants, tricyclic antidepressants) or decongestants, which may have serious drug interaction with hyoscine butylbromide
* suspected other alternative diagnoses (e.g. gut obstruction, biliary colic, pancreatitis, hepatitis or localized hepatobiliary infections, etc.)
* pregnancy or breast-feeding participants
* did not comprehend the Visual Analog Scale (VAS) evaluation

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khrongwong Musikatavorn, MD, Principal Investigator — Department of Medicine, Faculty of Medicine, Chulalongkorn University and King Chulalongkorn Memorial Hospital
Locations (1):
- Emergency Medicine Unit, King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand

REFERENCES:
- [Result] Musikatavorn K, Tansangngam P, Lumlertgul S, Komindr A. A randomized controlled trial of adding intravenous pantoprazole to conventional treatment for the immediate relief of dyspeptic pain. Am J Emerg Med. 2012 Nov;30(9):1737-42. doi: 10.1016/j.ajem.2012.02.001. Epub 2012 Mar 29. PMID 22463973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in January, 1 2011 and finished at the end October, 31 2011 in the Emergency Department of King Chulalongkorn Memorial Hospital
Pre-assignment Details: We analyzed the data for all enrolled patients with the intention-to-treat principles.
Period: Overall Study
Arm/Group | Conventional | Pantoprazole
Started | 44 | 43
Completed | 44 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional | Pantoprazole | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 4
  Between 18 and 65 years | 43 | 40 | 83
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.8 (8.1) | 29.4 (9.2) | 29.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 68
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  Thailand | 44 | 43 | 87
Pretreatment 100-millimeter visual analog scale (VAS) scores [Mean (Standard Deviation); unit: millimeters] — Self-marked pain scores on the 100-millimeter VAS lines were assessed by the patients before treatment. The minimal and maximal scores were between 0-100 millimeters. Good responders (good outcome) defined those had ≥ 50% decreases in post-treatment VAS compared with the pre-treatment evaluation and post-treatment scores ≤ 40 millimeters at the end of the study. Non-responders (worse outcome) defined those who had <50% decreases in post-treatment VAS compared with the pre-treatment evaluation or post-treatment scores > 40 millimeters at the end of the study.
  millimeters | 64 (13) | 64 (16) | 64 (14)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores on the 100-millimeter Visual Analog Scale (VAS) at 1 Hour After Treatment
Description: Post-treatment VAS will be consecutively measured every 15 minutes until 1 hour after treatment. Minimal and maximal VAS score of every measurement is 0 to 100 millimeters. VAS scores at 1 hour after treatment were the primary outcome measurement. The patients who had <50% decrement between pre- and 1-hour post-treatment VAS or post-treatment scores > 40 millimeters were defined as "Non-responders"(worse outcome). In the same way, those who had ≥ 50% decrement between pre- and 1-hour post-treatment VAS and post-treatment scores≤ 40 millimeters were defined as "Responders" (good outcome).
Time Frame: 1 hour after treatment
Population: All enrolled patients were analyzed with the intention-to-treat principles.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Conventional | Pantoprazole
Number analyzed (Participants) | 44 | 43
millimeter | 17 (24) | 19 (23)
Statistical Analysis 1: Comparison: Conventional vs Pantoprazole; Null hypothesis is that the treatment with pantoprazole arm is not different in immediate relief of acute, severe dyspeptic pain compared with conventional arm; Test type: Superiority or Other; p = 0.6, t-test, 2 sided; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-12.7 to 7.4], Standard Deviation 5.0

2. Secondary Outcome: Number of Participants in the Predefined "Responders"
Description: "Responders" define the participants who have ≥ 50% decrease in post-treatment pain scores compared with the pre-treatment evaluation and also have the post-treatment scores ≤ 40 at the end of the study.
Time Frame: pretreatment and 1 hour after treatment
Measure: Number; unit: participants
Arm/Group | Conventional | Pantoprazole
Number analyzed (Participants) | 44 | 43
participants | 36 | 32

3. Secondary Outcome: Number of Participants in the Predefined "Non-responders"
Description: "Non-responders" defined the participants who had < 50% decrease in post-treatment VAS compared with pre-treatment evaluation or post-treatment scores > 40 at the end of the study.
Time Frame: pretreatment and 1 hour after treatment
Measure: Number; unit: participants
Arm/Group | Conventional | Pantoprazole
Number analyzed (Participants) | 44 | 43
participants | 8 | 11

4. Secondary Outcome: Number of Participants With Adverse Effect
Description: The adverse effects include blurred vision, dry mouth, dizziness, headache, palpitation and diarrhea.
Time Frame: 1 hour after treatment
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants That Have Overall Satisfaction on the Treatment
Description: The satisfaction will be assessed by a simple, self-reported yes/no question.
Time Frame: 1 hour after treatment
Measure: Number; unit: participants
Arm/Group | Conventional | Pantoprazole
Number analyzed (Participants) | 44 | 43
participants | 34 | 34

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Conventional | Pantoprazole
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 31/44 | 30/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional (N=44) | Pantoprazole (N=43)
transient blurred vision (Eye disorders) | 22 (22) | 29 (29)
dry mouth (Gastrointestinal disorders) | 12 (12) | 6 (6)
dizziness (Nervous system disorders) | 3 (3) | 3 (3)
palpitation (Cardiac disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
1. This was a small, single-centered study. 2. Exaggerated self-evaluation of the patients' pain score and the physician's expectation of a "good outcome" may also have biased the report. 3. The short-term recurrence of the pain was not studied.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes